CLINICAL TRIAL: NCT07384663
Title: EFFICACY OF IV VERSUS ORAL IRON IN THE TREATMENT OF IRON DEFICIENCY ANEMIA DURING PREGNANCY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr Salaha Azam (Other)
Responsible Party: Sponsor-Investigator, Dr Salaha Azam, Principal Investigator, Doctors Hospital and Medical Centre Lahore
Organization: Doctors Hospital and Medical Centre Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 206
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Iron Deficiency Anaemia in Childbirth
Keywords: Anaemia; Iron Supplementation; Pregnancy
MeSH Terms: conditions — Anemia | interventions — ferric carboxymaltose; teferrol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A participants who were administered Intravenous Iron supplementation (Ferric carboxymaltose ) (Active Comparator): Treatment was initiated at the baseline visit. After baseline data was collected, women allocated to the IV iron group received a single dose of 500 mg Ferric carboxymaltose diluted in 100 mL 0.9% sodium chloride (or if pre-pregnancy body weight is < 50 kg the dose was 10 mg/kg based on pre-pregnancy body weight). Infusions were administered over approximately 20 min and participants were observed for adverse reactions during, and 30 min after, the end of the infusion. All randomized participants had scheduled follow-ups and outcome was assessed as per operational definition at 4th weeks. All data was collected on proforma.
  Interventions: Drug: Iron Carboxymaltose
- Group B participants who were administered Oral Iron Supplementation (polysaccharide iron complex) (Active Comparator): Women in the oral iron group received polysaccharide iron complex 150 mg capsule till 4 weeks. All randomized participants had scheduled follow-ups and outcome was assessed as per operational definition at 4th weeks. All data was collected on proforma.
  Interventions: Drug: Iron Polymaltose Complex

INTERVENTIONS:
Drug: Iron Carboxymaltose — Single dose of 500 mg Ferric carboxymaltose diluted in 100 mL 0.9% sodium chloride (or if pre-pregnancy body weight is < 50 kg the dose was 10 mg/kg based on pre-pregnancy body weight). Infusions was administered over approximately 20 min and participants were observed for adverse reactions during, and 30 min after, the end of the infusion.
  Arms: Group A participants who were administered Intravenous Iron supplementation (Ferric carboxymaltose )
Drug: Iron Polymaltose Complex — Polysaccharide iron complex 150 mg capsule was administered daily till 4 weeks
  Arms: Group B participants who were administered Oral Iron Supplementation (polysaccharide iron complex)

SUMMARY:
This study was planned to compare outcomes of IV versus oral iron in the treatment of iron deficiency anemia during pregnancy. This study was used to investigate the efficacy of two new formulations of iron both in IV and oral form with fewer side effects. We compared the efficacy of Intravenous Ferric Carboxymaltose with Oral polysaccharide iron complex. The better mode of treatment will be administered in future to treat this condition, that will surely improve the fetal and maternal outcome.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 -45 years;
* Second trimester (gestational age 14-21 weeks);
* Females having hemoglobin level of < 11 g/dL

Exclusion Criteria:

* Multiple pregnancies,
* A history of multiple allergies, known hypersensitivity to any of the excipients in the investigational drugs,
* Active infections
* Recent red blood cell (RBC) transfusion
* Thalassemia minor

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 112 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Blood Haemoglobin Levels | 4 weeks
  Non Anaemic Levels are labelled as (Hb ≥ 11.0 g/dL) at 4th week

CONTACTS AND LOCATIONS:
Locations (1):
- Doctors Hospital and Medical Centre Lahore, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No